CLINICAL TRIAL: NCT00294060
Title: Pacemaker Patient Profiling (P3) Study
Brief Title: P3: Pacemaker Patient Profiling Study
Status: Terminated | Type: Observational
Why Stopped: Preliminary analysis determined there was sufficient data to support objectives and allow early completion. The last patient visit occurred on November 6, 2007.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: P3 Study Team, Medtronic CRDM
Other Study IDs: 244
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-04

CONDITIONS: Bradycardia
Keywords: Pacemaker; Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The P3 Study is a United States post market study to gather data on clinical status, primary indications, device therapy choices, clinical management and outcomes for patients with implantable pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets Class I / Class II indications for pacing
* Patient implanted with one of the following market-approved single or dual chamber Medtronic devices: EnRhythm™, EnPulse®, Kappa® 700, Kappa® 900, Vitatron Clarity™, Vitatron Selection® AFm, Vitatron C-Series, Vitatron T-Series, or the AT500™ DDDR Pacing System

Exclusion Criteria:

* Patient is enrolled in a device or cardiovascular drug study that affects treatment and/or study device programming
* Patient whose life expectancy is less than two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2013 (Actual)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Kanagala, MD, Study Chair — Franciscan Skemp Healthcare
Locations (83):
- United States (83):
  - Birmingham, Alabama
  - Prescott, Arizona
  - Little Rock, Arkansas
  - Aliso Viejo, California
  - Anaheim, California
  - Arcadia, California
  - Escondido, California
  - Fountain Valley, California
  - La Mesa, California
  - Laguna Hills, California
  - Mission Viejo, California
  - Orange, California
  - Riverside, California
  - Tarzana, California
  - Whittier, California
  - Wildomar, California
  - Denver, Colorado
  - Fort Lauderdale, Florida
  - Lauderdale Lakes, Florida
  - Melbourne, Florida
  - Ocala, Florida
  - Sarasota, Florida
  - Vero Beach, Florida
  - Lawrenceville, Georgia
  - Idaho Falls, Idaho
  - Hinsdale, Illinois
  - Moline, Illinois
  - Hammond, Indiana
  - Terre Haute, Indiana
  - Hutchinson, Kansas
  - Edgewood, Kentucky
  - Owensboro, Kentucky
  - Lafayette, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Scarborough, Maine
  - Rockville, Maryland
  - Boston, Massachusetts
  - Cambridge, Massachusetts
  - Alpena, Michigan
  - Cleveland, Mississippi
  - Moberly, Missouri
  - Osage Beach, Missouri
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Kearney, Nebraska
  - Omaha, Nebraska
  - Bridgewater, New Jersey
  - Clifton, New Jersey
  - Elizabeth, New Jersey
  - Galloway, New Jersey
  - Elmira, New York
  - Huntington, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Cleveland Heights, Ohio
  - Columbus, Ohio
  - Dublin, Ohio
  - Kettering, Ohio
  - Lima, Ohio
  - Lorain, Ohio
  - Mayfield Heights, Ohio
  - Middleburg Heights, Ohio
  - Zanesville, Ohio
  - Tulsa, Oklahoma
  - Wakefield, Rhode Island
  - Greenville, South Carolina
  - Sumter, South Carolina
  - Austin, Texas
  - Beaumont, Texas
  - Houston, Texas
  - Humble, Texas
  - Lubbock, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Victoria, Texas
  - Wichita Falls, Texas
  - La Crosse, Wisconsin
  - Waukesha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in the study from March 2004 through April 2006.
Pre-assignment Details: Only patients who received an approved study device were enrolled in the registry.
Groups:
- Pacing Patients: Patients implanted with a pacemaker.
Period: Overall Study
Arm/Group | Pacing Patients
Started | 2013
Completed | 840
Not Completed | 1173
Not completed — Death | 225
Not completed — Other | 59
Not completed — Lost to Follow-up | 55
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 797
Not completed — Medical condition | 3
Not completed — Device explanted/not replaced | 23

BASELINE CHARACTERISTICS:
Arm/Group | Pacing Patients
Number analyzed (Participants) | 2013
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 266
  >=65 years | 1747
Age Continuous [Mean (Standard Deviation); unit: years] | 76.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 996
  Male | 1017
Region of Enrollment [Number; unit: participants]
  United States | 2013

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dual Chamber Devices
Description: Pacemaker device choice characterized by the number of patients with dual chamber devices
Time Frame: at original implant
Measure: Number; unit: Participants with dual chamber devices
Arm/Group | Pacing Patients
Number analyzed (Participants) | 2013
Participants with dual chamber devices | 1684

2. Primary Outcome: Days Hospitalized
Description: Healthcare utilization clinical outcome characterized by number of days hospitalized in the first year
Time Frame: implant to one year
Population: Patients with a twelve-month follow-up visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: average days hospitalized
Arm/Group | Pacing Patients
Number analyzed (Participants) | 1211
average days hospitalized | 0.054 (2.35)

3. Primary Outcome: Multiple In-clinic Visits
Description: Follow-up practice pattern assessed by the number of patients with a dual chamber device that had two or more routine pacemaker in-clinic visits with a device interrogation
Time Frame: implant to one year
Population: Only those patients with a dual chamber device completing 12 months of follow-up were included in this analysis.
Measure: Number; unit: participants with 2 or more visits
Arm/Group | Pacing Patients
Number analyzed (Participants) | 1459
participants with 2 or more visits | 768

ADVERSE EVENTS:
Time Frame: Adverse events were not collected in the P3 Study. The products used in the study are market approved and were used within the indications for use as indicated in the product labeling.
Description: Centers were instructed to report Unanticipated Adverse Device Events (UADE) in the same manner as required for any commercially available device, that is, through the Medical Device Reporting (MDR) processes and in accordance with any reporting requirements required by their IRB.
Arm/Group | Pacing Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Characterization of objectives also encompassed 8 device features (Capture Management, MVP, APP, ARS, PMOP, Rate Response, Mode Switch, Sinus Preference) and 10 additional clinical outcomes. More information is available through the point of contact.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators to publish study results per the publication plan/protocol following Medtronic's review to determine whether confidential information ("CI") is disclosed. Any such CI is deleted prior to publication/presentation. Medtronic may not censor/interfere with the publication except as described. Investigators may not publish any single-site publications until the main multi-site study publication has occurred.